CLINICAL TRIAL: NCT00246961
Title: Arimidex: Reason for and Effect of Change From Tamoxifen
Brief Title: Arimidex Observational: Reason for and Effect of Change From Tamoxifen
Acronym: ARREST
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: D5392NL0002; ARREST
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer
Keywords: Adjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyse the effect on quality of life after 3 months of treatment after changing adjuvant therapy from tamoxifen to Arimidex.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Hormone sensitive breast cancer
* Patient uses tamoxifen or has stopped taking tamoxifen less than 7 days ago

Exclusion Criteria:

* Visceral metastases
* Patients with signs of progression at the moment of changing therapy
* Patients who have used other endocrine treatments for breast cancer besides tamoxifen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca The Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (33):
- Netherlands (33):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Antwerpen
  - Research Site, Apeldoorn
  - Research Site, Bergen op Zoom
  - Research Site, Boxmeer
  - Research Site, Breda
  - Research Site, Doetinchem
  - Research SIte, Dordrecht
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Flushing
  - Research Site, Geldrop
  - Research Site, Groningen
  - Research Site, Harderwijk
  - Research Site, Helmond
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Leiden
  - Research Site, Oosterhout
  - Research Site, Purmerend
  - Research Site, Roermond
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Venray
  - Research Site, Winterswijk
  - Research Site, Zoetermeer
  - Research Site, Zutphen